CLINICAL TRIAL: NCT06918587
Title: Open Label Randomized Two Treatment Two Sequence Two Period Crossover Single Dose Pharmacokinetic Immunogenicity and Safety Study of Pegfilgrastim Comparing TPI-120 Prefilled Syringe With on Body Injector 6mg as Test Product (T) Manufactured by Kashiv Biosiciences LLC, USA With Fylnetra Prefilled Syringe 6mg as Reference Product (R) Manufactured by Kashiv Biosciences LLC, USA Administered Through Subcutaneous Route in Normal Healthy Adult (Males and Females ) Human Subjects Under Fasting Condition
Brief Title: Open Label Randomized Comparative Crossover Pharmacokinetic and Immunogenicity Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kashiv BioSciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TPI-120 with On Body Injector
Record Dates: First submitted 2025-01-31; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Febrile Neutropenia
Keywords: pegfilgratim; on body injector
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: An Open label, randomized, single-dose, two sequences, two-period , two-arm crossover comparative Pharmacokinetic, immunogenicity and safety study under fasting conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Product TPI-120 with On body Injector 6 mg (Experimental): On body injector
  Interventions: Device: TPI-120 with On body injector
- Fylnetra (Active Comparator): Fylnetra 6mg
  Interventions: Drug: Fylntera

INTERVENTIONS:
Device: TPI-120 with On body injector — 6mg Subcutaneous injection
  Arms: Test Product TPI-120 with On body Injector 6 mg
Drug: Fylntera — 6mg subcutaneous
  Arms: Fylnetra

SUMMARY:
The Goal of these study is to evaluate and To compare the pharmacokinetics (PK) of the Test product (T) getting administered through prefilled syringe with on-body injector with Reference product as prefilled syringe following a single 6 mg dose administered through subcutaneous route in healthy adult Human subjects.

Subjects safety and immunogenicity will also be evaluated during these study as follows Safety - monitoring the adverse events , vitals signs, ECG, laboratory parameters, and injection site assessment.

Immunogenicity assessment- detection of ADA (Anti-PEG antibody levels ) and Nab (Neutralizing antibodies) will be done pre-dose and post dose on day 15 of each period.

ELIGIBILITY:
Inclusion Criteria:

1. - Subjects are physically and mentally healthy adults aged between 18 and 50 years (both inclusive) at screening.

2.Subject's weight within normal range according to normal values for Body Mass Index (18.5 to 30.0 kg/m2) (both inclusive) with minimum of 50 kg weight at screening.

3.The findings of the subject are within the range of clinical acceptability in medical history, medication history, clinical examination, and laboratory examinations "other than RBC indices (MCH, MCV and MCHC) and hemoglobin" are within "normal ranges" or abnormalities considered insignificant and justified by the principal/clinical sub- Investigator at screening.

4.The subject results of all RBC indices (MCH, MCV and MCHC) and hemoglobin are within normal range or ± 5% of medical lab reference range at screening.

5.The subject's kidney function tests (Serum Creatinine, Potassium, Sodium) are within the medical lab reference range, and kidney function tests (urea, and chloride) are considered clinically acceptable as per the investigator judgment at screening. If creatinine is below the lower normal limit while the other parameters are normal, it will be considered as clinically not significant unless otherwise judged by the investigator.

The subject's Liver function tests (AST, ALT, GGT, and total bilirubin) results are within the medical lab reference ranges and liver function tests (Alkaline phosphatase, total protein, and albumin) are considered clinically acceptable as per PI / SI judgment at screening.

7.The subject's Cholesterol level is considered clinically acceptable as per PI / SI judgment at screening.

8.The subject is fasting for at least 12 hrs before giving the samples required for clinical laboratory examinations as checked at screening .

9.Subject having vital signs parameters (blood pressure, body temperature, pulse rate and respiratory rate) are within the following ranges at screening, and on admission day (before admission) of period I: Blood Pressure: Systolic: (90- 140) mmHg, Diastolic: (60-90) mmHg Body Temperature: (36.1 - 37.2) ºC Pulse rate: 60 to 100 beat per minute. Respiratory rate: 12-18 bpm. 10.Subject complies with Injection site evaluation at screening and on admission day (before admission) of period I.

11.The subject has a normal ECG (12 leads) as per the investigator judgement, at screening and on admission day (before admission) of period I.

12.The subject has normal abdominal ultrasonography (no signs of spleen rupture or splenomegaly) as checked at screening 13.The subject has clinically acceptable chest x-ray (PA view) as per the investigator judgment as checked at screening.

14.The subject has having negative urine screen for drugs of abuse (amphetamine, barbiturates, benzodiazepines, cocaine, opiates, marijuana, methadone, methamphetamine, phencyclidine, and Tricyclic antidepressants) at screening and on admission day (before admission) of period I .

15.The subject has negative alcohol test at screening and on admission day (before admission) of period I.

16.The subject (available for entire study duration) is willing to adhere to the protocol requirements and to provide signed informed consent (by applying his / her signature or fingerprint) as confirmed at screening and on admission day (before admission) of period I.

Females of non-childbearing potential must have undergone sterilization procedures, at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status 18.For Female Subjects "who have the potential to become pregnant":

* The subject has negative serum pregnancy test at screening and on admission day (before admission) of period I.
* Female of child bearing potential agrees to practice for the duration of the study an acceptable method of birth control as judged by the investigator(s), such as intrauterine device (IUD), abstinence or double barrier contraception, i.e., condom + diaphragm, condom + spermicidal or foam prior to the start of the study and through the study and for 30 days after last dosing in study as checked at screening and on admission day (before admission) of period I.

  19.The male subject agrees, at screening and on admission day (before admission) of period I, to use a condom for the duration of the study, and for 30 days after last dosing in study if:He is engaged in sexual activity with a woman of childbearing potential.
* A condom is required along with another medically acceptable contraceptive method. Medically acceptable methods of contraception include non-hormonal intrauterine device or double barrier method (condom with foam or vaginal spermicidal suppository, diaphragm with spermicide).
* Not to donate sperms during the study and for 30 days after last dosing in study

Exclusion Criteria:

Subjects will be excluded from the study, if they meet any one of the following criteria:

1. The subject has history of allergy or hypersensitivity to study drug or adhesive material or related class of drugs or to the inactive ingredients (acetate/acetic acid, polysorbate 20, or sorbitol) of the test and reference formulation as checked at screening.
2. The subject has history or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological disease, or disorder as checked at screening or on admission day (before admission) of period I.
3. The subject has an evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of the consent to participation in the study or limit the ability to comply with the protocol requirements, as determined by the principal investigator/clinical sub-investigator at screening or on admission day (before admission) of period I.
4. The subject has a clinically significant history of skin disorders, including psoriasis or any clinically significant skin abnormality at injection site as checked at screening or on admission day (before admission) of period I.
5. The subject has a history of any of the following, as checked at screening: Autoimmune disease.

   * Splenic Rupture or Splenomegaly.
   * Acute respiratory distress syndrome
   * Sickle Cell Disorders
   * Glomerulonephritis
   * Leukocytosis
   * Thrombocytopenia
   * Capillary Leak Syndrome
   * History of cancer; or malignant Cells.
   * Aortitis
   * History of pulmonary infiltrate or pneumonia (radiologically confirmed) within 6 months prior to initial dosing.
   * Any past exposure to recombinant human G-CSF products and/or a known history of prior treatment with blood-cell colony stimulating factors, interleukins or interferons.

History or presence of asthma, urticaria or other significant allergic reactions as checked at screening.

7.History or presence of significant gastric and/or duodenal ulceration as checked at screening.

8.The subject has received any vaccination (including influenza) within 60 days prior to first dosing as checked at screening.

9.The subject used any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month prior to dosing of Period I as checked at screening or on admission day (before admission) of period I.

10.The subject is a moderate smoker (more than 10 cigarettes per day) as checked at screening or on admission day (before admission) of period I 11.History or presence of drug abuse in the past one year as checked at screening.

12.History or presence of alcohol abuse in the past one year [alcohol abuse will be >14 drinks per week (1 drink = 360 mL beer, 150 mL wine, or 45 mL hard liquor)] as checked at screening.

13.Difficulty with donating blood as checked at screening or on admission day (before admission) of period I.

14.Use of any prescribed medication or OTC medication including vitamins and herbal remedies during last 14 days prior to dosing in period I as checked at screening or on admission day (before admission) of period I.

15.Major illness or hospitalization within past 3 months as checked at screening or on admission day (before admission) of period I.

16.Volunteer/s who have donated 1 unit blood (≥ 300 mL) or participated in a clinical study involving blood sampling within 80 days prior to the first dose of the study drug as checked at screening or on admission day (before admission) of period I.

17.Consumption of grapefruit juice, caffeine, poppy seeds, within 72 hours prior to dosing and other xanthine-containing products, tobacco containing products or any alcoholic products within 48 hours prior to dosing as checked on admission day (before admission) of period I .

18.Positive test for one or more: HIV, Hepatitis B and Hepatitis C at screening.

19.History or presence of significant easy bruising or bleeding as checked at screening.

History or presence of significant recent trauma as checked at screening. 21.Female volunteer who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing as checked at screening or on admission day (before admission) of period I.

22.Female subjects who are currently breast feeding as checked at screening or on admission day (before admission) of period I.

23.Pregnant female volunteers as checked at screening or on admission day (before admission) of period I.

24.Known allergies to acrylics (as the on-body injector uses acrylic adhesive) as checked at screening or on admission day (before admission) of period I.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pharmackinetic Outcomes | Blood samples (5.0 mL) will be collected at pre-dose (00.00 hr) in the morning on dosing day (day 1) within 01.00 hour prior to dosing and at 00.33, 00.50, 00.75, 01.00, 02.00, 04.00, 06.00, 08.00, 10.00, 12.00, 14.00, 16.00, 20.00, 24.00 (day 2), 36.00,
  Primary PK parameters: Cmax
Pharmacokinetic outcomes | Blood samples (5.0 mL) will be collected at pre-dose (00.00 hr) in the morning of dosing day (day 1) within 01.00 hour prior to dosing and at 00.33, 00.50, 00.75, 01.00, 02.00, 04.00, 06.00, 08.00, 10.00, 12.00,14.00, 16.00, 20.00, 24.00 (day 2), 36.00,
  AUC0-t

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pallav Bharpoda, MBBS PGDCR, Study Director — Kashiv biosciences
Locations (1):
- Not Disclosed, Jordan, Jordan